CLINICAL TRIAL: NCT04624477
Title: Active Surveillance or Surgery for Primary Management of Very Low Risk Papillary Thyroid Cancer: How Often Are the Long-term Disease Management Goals Achieved?
Brief Title: Active Surveillance and Surgery Outcomes in Low Risk Papillary Thyroid Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of British Columbia (Other); University of Calgary (Other); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other); McMaster University (Other); CHU de Quebec-Universite Laval (Other); Dalhousie University (Other); Canadian Cancer Society (CCS) (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 20-5102
Record Dates: First submitted 2020-10-27; First posted 2020-11-10 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Papillary Thyroid Cancer; Papillary Thyroid Carcinoma; Papillary Microcarcinoma of the Thyroid
Keywords: papillary thyroid cancer; papillary thyroid carcinoma; thyroid cancer; thyroid carcinoma; thyroid microcarcinoma; low risk thyroid cancer; active surveillance; thyroidectomy
MeSH Terms: conditions — Thyroid Cancer, Papillary; Papillary Thyroid Microcarcinoma; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active Surveillance: Patients under active surveillance choose to not have immediate thyroid surgery. Patients are closely monitored with respect to clinical status, ultrasound imaging, biochemical indices (thyroid function, thyroglobulin, and thyroglobulin antibodies) and any thyroid cancer-related treatments (if received). Active surveillance is conducted at a participating study site. Criteria defining disease progression are established, and if such criteria are met, thyroid surgery is recommended to the patient. However, patients are free to choose to have thyroid surgery at any time, in the absence of disease progression. Thyroid cancer clinical and treatment outcomes are tracked by the study team.
- Immediate Thyroid Surgery (total or partial thyroidectomy): Patients who choose surgery, undergo thyroidectomy, as per current standards of care, by a surgeon of their choice in an institution of their choice. The treating surgeon, in discussion with the patient, will choose the extent of thyroid surgery that may be appropriate for the individual case. Post-surgical follow-up is per the discretion of the treating surgeon, endocrinologist, or other healthcare providers involved in the patient's thyroid cancer care. Thyroid cancer clinical and treatment outcomes are tracked by the study team.

SUMMARY:
This is a prospective, observational, multi-center study examining the long-term outcomes of patients with small, low risk papillary thyroid cancer who offered the choice of active surveillance (close follow-up to monitor for potential disease progression) or immediate surgery.

DETAILED DESCRIPTION:
This is a prospective, observational multi-center study, building on an initial single-centre study from Toronto, Canada (ClinicalTrials.gov Identifier: NCT03271892). Adult patients with small, low-risk papillary thyroid cancer may choose either active surveillance (close follow-up with the intention of surgery if the disease progresses or if the patient changes their mind and wants surgery) or immediate thyroid surgery (thyroidectomy). Patients who choose active surveillance are clinically followed at the participating study centre and those who choose surgery, receive usual care from their treating surgeon and/or other thyroid cancer specialists.

Thyroid cancer clinical and treatment outcomes are tracked (by medical record review) at least yearly for up to 10 years after enrollment. Patients are also asked to complete study questionnaires (patient reported outcomes) yearly for up to 5 years.

The underlying assumption in the study is that since patients' disease management goals differ for individuals choosing active surveillance and those choosing surgery, 'successful' disease management is defined differently for these patient groups. For patients choosing active surveillance, successful disease management may be defined by avoiding thyroid surgery for thyroid cancer progression (i.e. thyroid cancer that has grown or spread to other tissues). For patients choosing surgery, the ultimate goal is cure of the thyroid cancer (i.e. no thyroid cancer detected at long-term follow-up).

The primary analysis in this study is a description of how often patients' initial disease management goals are not achieved at long-term follow-up. For this study, 'failure' of disease management is defined as follows: a) in active surveillance group - surgery for disease progression, and b) in the immediate surgery group - requiring additional treatment for persistent or recurrent thyroid cancer (i.e. thyroid cancer that is detected and treated in follow-up). Thyroid cancer clinical and treatment outcomes as well as patient questionnaire outcomes will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older.
* Newly diagnosed previously surgically untreated papillary thyroid cancer (PTC) or suspicious for PTC on fine needle aspiration biopsy of the thyroid. PTC must be < 2 cm in maximal diameter on thyroid ultrasound.
* The absence of metastatic cervical lymphadenopathy or gross extrathyroidal extension of PTC, as confirmed on neck ultrasound imaging.
* The absence of other current absolute indication for thyroid or parathyroid surgery (e.g. severe hyperthyroidism that cannot be controlled medically, large goitre with severe compressive symptoms, or primary hyperthyroidism meeting surgical criteria).

Exclusion Criteria:

* Metastatic thyroid cancer (lymph nodes or distant).
* History of prior thyroid surgery for any indication.
* The primary PTC being on the trachea or immediately adjacent to the recurrent laryngeal nerve, and with progression would be deemed to be at high risk of growth into these critical structures.
* Clinical signs, imaging, or laryngoscopy findings suggestive of locally advanced thyroid cancer (i.e. vocal cord paralysis due to the thyroid cancer or any clinical or radiographic signs of extrathyroidal invasion into adjacent structures such as the strap muscles of the neck, trachea or esophagus).
* Known/suspected poorly differentiated or non-papillary thyroid cancer.
* Medically unfit for surgery due to severe co-morbidity. Severe comorbidity may include another active malignancy with limited life expectancy of < 1 year).
* Pregnancy at the time of study enrollment.
* Unable/unwilling to provide informed consent for the study or comply with study follow-up procedures due to current active physical limitations/medical co-morbidity, cognitive, or psychiatric impairment substance abuse, or other reasons.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults (aged 18 years of age or older) with small (< 2cm maximal diameter) low risk papillary thyroid cancer that is confined to the thyroid (with no evidence of metastatic disease, no extrathyroidal extension, which is not in a location that is of high risk for invasion of the trachea or recurrent laryngeal nerve).
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants in the Active Surveillance Group who Experience 'Failure' of Active Surveillance Disease Management | Through study completion, an estimated average of 3 years
  'Failure' of Active Surveillance Disease Management is defined as: surgery for the indication of thyroid cancer that has progressed during study monitoring. Thyroid cancer disease progression under active surveillance includes: a) thyroid cancer enlargement > 3mm in largest dimension, b) thyroid cancer growth in a location that is concerning (e.g. extension outside of the thyroid, concerning proximity to critical structures such as the trachea or recurrent laryngeal nerve), or c) development of metastatic disease (in lymph nodes or distant organs). The specific type of disease progression will be reported.
Number of Participants in the Surgical Group who Experience 'Failure' of Surgical Disease Management | Through study completion, an estimated average of 3 years
  For patients who choose immediate surgery for management of thyroid cancer, the intent of surgery is curative. Thus, 'failure' of surgical disease management is defined by receiving additional treatment for structural thyroid cancer detected at follow-up (i.e. treatment of thyroid cancer detected on imaging or biopsy during follow-up). Additional thyroid cancer treatment may include additional surgery, radioactive iodine, ethanol ablation of lymph nodes, or external beam radiation treatment. The specific treatment used for recurrent or persistent thyroid cancer and the indication for the treatment will be reported.

SECONDARY OUTCOMES:
Number of Participants in Respective Thyroid Cancer Disease Status Categories at Last Follow-up | Through study completion, an estimated average of 3 years
  The category of thyroid cancer disease status at last follow-up is recorded at least yearly. For patients in the active surveillance arm, disease status categories include: a) alive with no disease progression, b) alive with cross-over to surgery (with indication for surgery, including disease progression or other reason), c) death due to thyroid cancer, or d) death from any cause. For surgical patients and patients who crossed over to surgery from active surveillance, post-surgical disease status categories include: a) alive with no evidence of thyroid cancer structural disease at last follow-up (e.g.. no evidence of thyroid cancer on imaging or biopsy), b) alive with evidence of thyroid cancer structural disease present at last follow-up (i.e. evidence of thyroid cancer on imaging or biopsy), c) death due to thyroid cancer, or d) death from any cause.
Number of Participants in the Active Surveillance Group who Undergo Thyroidectomy During Follow-up | Through study completion, an estimated average of 3 years
  The number of participants in the active surveillance group who cross over to thyroidectomy during follow-up (with the specific indication for the thyroidectomy and type of thyroid surgery) will be reported.
Number of Participants who Experience Long-term Complications of Thyroid Surgery | Through study completion, an estimated average of 3 years
  For patients who undergo thyroidectomy during the study, the presence of long-term surgical complications (> 1 year after initial completion of surgery) will be reported. Specific surgical complications that will be tracked include: a) hypoparathyroidism (requiring prescription treatment), or b) recurrent laryngeal nerve injury.
Description of Quality of Life (Thyroid Cancer-specific) | Through study completion, an estimated average of 3 years
  EORTC QLQ-THY34 (all respective scales). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. All of the scales and single item measures range in score from 0 to 100. A high score for the symptom scales and single items indicates a worse outcome, whereas a high score for the Social Support scale represents a high level of functioning.
Description of Quality of Life (Cancer-specific) | Through study completion, an estimated average of 3 years
  EORTC QLQ-C30 (all respective scales). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high / healthy level of functioning (better outcome), a high score for the global health status /quality of life represents a better outcome, but a high score for a symptom scale / item represents a worse outcome.
Measure of Anxiety | Through study completion, an estimated average of 3 years
  Generalized Anxiety Disorder Screener questionnaire (minimum score 0, maximum score 21, where a higher score indicates a worse outcome)
Measure of Survivor Concerns | Through study completion, an estimated average of 3 years
  Assessment of Survivor Concerns questionnaire (Cancer Worry Subscale - minimum score 3, maximum score 12, where a higher score indicates a worse outcome and General Health Worry Subscale - minimum score 2, maximum score 8, where a higher score indicates a worse outcome)
Measure of Decision Regret (relating to the original decision to undergo active surveillance or thyroid surgery). | Through study completion, an estimated average of 3 years
  Decision Regret Scale (minimum score 0, maximum score 100, where a higher number indicates a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Sawka, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (8):
- Canada (8):
  - University of Calgary, Cumming School of Medicine, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Nova Scotia Health, Halifax, Nova Scotia
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Lawson Health Research Institute, London, Ontario
  - University Health Network, Toronto, Ontario
  - Division chirurgie ORL et cervico-faciale, Montreal, Quebec
  - CHU de Québec - Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No
Individual sites will have access to individual participant data from their own site.

REFERENCES:
- [Background] Sawka AM, Ghai S, Tomlinson G, Baxter NN, Corsten M, Imran SA, Bissada E, Lebouef R, Audet N, Brassard M, Zhang H, Gupta M, Nichols AC, Morrison D, Johnson-Obeski S, Prisman E, Anderson D, Chandarana SP, Ghaznavi S, Jones J, Gafni A, Matelski JJ, Xu W, Goldstein DP; Canadian Thyroid Cancer Active Surveillance Study Group. A Protocol for a Pan-Canadian Prospective Observational Study on Active Surveillance or Surgery for Very Low Risk Papillary Thyroid Cancer. Front Endocrinol (Lausanne). 2021 Jun 10;12:686996. doi: 10.3389/fendo.2021.686996. eCollection 2021. PMID 34194396